CLINICAL TRIAL: NCT07025070
Title: The Link Between Strength and Endurance Training and Brain Health in Healthy Adults: A Comparative Study of Former Professional Athletes and Sedentary Individuals
Brief Title: The Link Between Physical Activity and Brain Health in Healthy Adults
Acronym: MINA
Status: Recruiting | Type: Observational
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, Songxin Tang, Principal Investigator, Technical University of Madrid
Other Study IDs: MINAEPSLRE-MMGG-DATOS-20240219; S2022/BMD-7236 (Other Grant/Funding Number: Research groups of the Community of Madrid in Biomedicine)
Record Dates: First submitted 2025-05-27; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Inactivity; Preventive Therapy
Keywords: physical activity
MeSH Terms: conditions — Alzheimer Disease; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Detection of mutated genes associated with early-onset Alzheimer's disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ex-athletes and continue to exercise regularly
- Sedentary individuals

SUMMARY:
The goal of this observational study is to investigate the cross-sectional relationship between physical activity and brain health from a multiscale approach (neuropsychology, neuroimaging, peripheral biomarkers and genetics) in former athletes and sedentary individuals. The main question it aims to answer is:

Do former athletes have better brain structure than sedentary people? Evaluating the differences in neurodegenerative processes between competitive training and sedentary and inactivity.

ELIGIBILITY:
Inclusion Criteria:

* Group A: ex-athletes and continue to perform regular physical exercise (minimum 3 days/week of moderate-vigorous intensity).
* Group B: sedentary individuals, (i.e., perform <150 min of moderate intensity exercise per week or IPAQ score<600 MET min/week).
* In both groups (A and B) the conditions of physical exercise or sedentary lifestyle must have been maintained for at least 6 months prior to the evaluations.
* Not having a history of neurological or psychiatric disorder or suffering from a serious medical condition

Exclusion Criteria:

* Medical conditions that have a high risk of associated cognitive symptoms.
* Severe head injury with loss of consciousness within the previous 5 years.
* Alcoholism (>3 alcoholic drinks per day).
* Chronic use of anxiolytics, neuroleptics, narcotics, anticonvulsants, or sedative hypnotics.
* Hearing or visual impairment that would preclude testing
* History of neurological disease with clinically relevant impact on cognition (e.g. cerebrovascular disease).
* Incidental structural brain findings with impact on cognitive impairment or survival (e.g., malignant brain tumor).
* Presence of severe systemic disease (e.g., cancer under treatment).
* Consumption of anabolic substances.
* Problems understanding spoken or written Spanish.
* Those with pacemakers or metallic implants that may interfere with the MRI.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Region of Madrid
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Concentration of brain-derived neurotrophic factor (BDNF) in plasma (pg/mL) | Baseline
  Measured with ELISA kit (e.g., R&D Systems, Cat. #DY248). Higher BDNF reflects greater neurotrophic support.
Concentration of total tau protein in plasma (pg/mL) | Baseline
  Assayed by high-sensitivity ELISA (e.g., Cusabio, Cat. #CSB-E13913h). Greater tau concentration indicates increased axonal injury or neurodegeneration.
Hippocampal volume measured by high-resolution 3 T T1-weighted MRI (mm³) | Baseline
  Volume extracted with FreeSurfer; Larger values indicate greater hippocampal integrity
Resting-state functional connectivity between primary motor cortex and supplementary motor area measured by 3 T fMRI (Fisher-Z) | Baseline
  Fisher-Z transformed correlation computed with CONN; Higher values indicate stronger connectivity
Digit Span Forward maximum span length (digits) | Baseline
  Attention assessed with Wechsler Adult Intelligence Scale-IV Digit Span Forward subtest; Maximum correctly repeated digit sequence recorded. Higher scores indicate better attention/short-term memory capacity.
Trail Making Test Part A completion time (seconds) | Baseline
  Visual attention and processing speed measured by TMT-A; time to connect 25 numbers in ascending order recorded. Shorter times indicate better performance.
Digit Span Backward maximum span length (digits) | Baseline
  Working memory measured with WAIS-IV Digit Span Backward; Longest correctly repeated backward sequence recorded. Higher scores indicate better working memory.
Trail Making Test Part B completion time (seconds) | Baseline
  Executive function (set-shifting) assessed by TMT-B; Time to alternately connect numbers and letters recorded. Shorter times indicate better executive control.
Verbal fluency (F-A-S) total words in 60 s (count) | Baseline
  Phonemic fluency tested with Controlled Oral Word Association Test (letters F, A, S, 60 s each); total correct words across three letters. Higher counts indicate better executive retrieval fluency.
Stroop Color-Word interference score (seconds) | Baseline
  Inhibition assessed with Golden Stroop test; The count of completions within 45 seconds is recorded. Lower times reflect better inhibitory control.
Montreal Cognitive Assessment (MoCA) total score (0 - 30 points) | Baseline
  10-minute screening of global cognition covering memory, attention, language, visuospatial, and executive domains. Values ≥ 26 are considered normal. Higher scores indicate better cognition.
Number of participants carrying at least one APOE ε4 allele (count of participants) | Baseline
  Genomic DNA isolated from EDTA whole blood; APOE genotyping by TaqMan SNP assays rs429358 and rs7412. Any ε4-containing genotype (ε2/ε4, ε3/ε4, ε4/ε4) classified as "ε4 carrier". Higher counts = higher ε4 prevalence.

SECONDARY OUTCOMES:
Maximal oxygen uptake (VO₂max) measured by CPET with ramp protocol on treadmill (mL·kg-¹·min-¹) | Baseline
  Cardiopulmonary exercise test performed on treadmill using Ramp incremental ramp. Breath-by-breath gas exchange collected via metabolic cart. VO₂max defined as the highest 30-s average during the test; Higher values indicate better cardiorespiratory fitness.
Mean daily minutes of moderate-to-vigorous physical activity measured by ActiGraph wGT3X-BT accelerometer over 7 days (min/day) | Baseline
  Device worn on non-dominant wrist 24 h/day for 7 consecutive days. Raw data (100 Hz) processed in ActiLife with 10 s epochs; Freedson adult cut-points ≥ 1 952 counts·min-¹ define MVPA. Higher values indicate greater physical activity.
Body mass index (BMI) calculated from weight and stadiometer-measured height (kg/m²) | Baseline
  Height measured to 0.1 cm with height measuring rod. Weight obtained from InBody system. BMI = weight ÷ height². Higher BMI indicates greater overall adiposity.
Peak force of mid-thigh-pull test measured by portable force dynamometer (N) | Baseline
  Participants perform two maximal isometric mid-thigh pulls on calibrated dynamometer with 60 s rest. The higher of two trials recorded as peak force. Greater values indicate stronger lower-limb strength.
Handgrip strength measured by grip dynamometer (kg) | Baseline
  Standing posture, shoulder neutral, elbow extended. Two maximal squeezes per hand with dynamometer; 30 s rest between trials. Best value used for analysis. Higher values reflect greater grip strength.
Timed Up-and-Go (TUG) test completion time (seconds) | Baseline
  Participants stand up from a 45-cm chair, walk 3 m, turn, return, and sit; time recorded by timers. Two trials with 1 min rest; Shorter time retained. Lower times represent better agility.
Balance stability and speed score measured by TANITA force platform (unitless) | Baseline
  Balance and speed assessed on TANITA analyzer in eyes-open seated posture; Stand-up as fast as possible when signaled, repeat 3 times to get an optimal value; Manufacturer's composite stability index automatically computed (range 0-100). One 30-s trial; higher scores denote better balance.
Percentage body fat measured by multifrequency bioimpedance analyzer InBody system (%) | Baseline
  Participants barefoot, InBody 770 provides whole-body fat percentage derived from segmental impedance; Higher values denote greater adiposity.
Skeletal muscle mass measured by multifrequency bioimpedance analyzer InBody system (kg) | Baseline
  Analyzer outputs total skeletal muscle mass. Greater values indicate higher muscularity.
Waist circumference measured by flexible tape at midpoint between lowest rib and iliac crest (cm) | Baseline
  Measured at end-expiration; two readings within 1 cm averaged. Larger values indicate central adiposity.
Hip circumference measured by flexible tape at level of greater trochanters (cm) | Baseline
  Two readings averaged; used with waist girth to compute waist-to-hip ratio.
Serum triglycerides measured by enzymatic colorimetric assay (mg/dL) | Baseline
  Fasting venous blood; triglycerides quantified on chemistry analyzer with glycerol phosphate oxidase method. Higher values indicate greater dyslipidemia risk.
Serum total cholesterol measured by enzymatic colorimetric assay (mg/dL) | Baseline
  Chemistry analyzer; Cholesterol esterase/oxidase method. Higher levels indicate increased cardiovascular risk.
Serum high-density lipoprotein (HDL) cholesterol measured by enzymatic assay (mg/dL) | Baseline
  Selective detergent method. Higher HDL is considered protective.
Serum low-density lipoprotein (LDL) cholesterol calculated by Friedewald formula (mg/dL) | Baseline
  LDL-C = total-C - HDL-C - (triglycerides ÷ 5). Higher LDL indicates greater atherogenic risk.
Serum 25-hydroxyvitamin D concentration measured by chemiluminescent immunoassay (ng/mL) | Baseline
  Serum 25-hydroxyvitamin D concentration measured by chemiluminescent immunoassay (ng/mL)
Mean daily sedentary time measured by ActiGraph wGT3X-BT accelerometer over 7 days (min/day) | Baseline
  Sedentary time defined as < 100 counts·min-¹ in vector-magnitudes; summed across valid waking wear days (≥ 10 h/day). Larger values denote more sedentary lifestyle.
Mean nightly sleep duration measured by ActiGraph wGT3X-BT over 7 nights (hours/night) | Baseline
  Sleep/wake scored with Cole-Kripke algorithm; average total sleep time across nights with ≥ 160 min valid sleep. Longer duration indicates better sleep quantity.
Total physical activity measured by International Physical Activity Questionnaire - Long Form (MET·min/week) | Baseline
  Four IPAQ domains are summed; for each activity, minutes are multiplied by the corresponding MET value and then summed. Higher values indicate greater total energy expenditure.
Mediterranean Diet Adherence Score measured by 14-item Mediterranean Diet Adherence Screener (0 - 14 points) | Baseline
  Each of the 14 items is scored 0 or 1 and summed (total 0-14). A score ≥ 9 is considered high adherence. Higher scores indicate greater adherence to the Mediterranean dietary pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Activity and Sports Sciences (INEF), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, the investigators have not yet decided whether our IPD will be shared. Data sharing policies and procedures are still under discussion within our research group and institution. Further consideration will be given to ethical requirements, participant privacy, and potential future analyses before making a final decision.

REFERENCES:
- See also: Related Info — https://imfine.com.es/